CLINICAL TRIAL: NCT04816084
Title: SERUR : Etude sérologique COVID-19 (Anti-SARS CoV 2) du Personnel de l'Université de Reims Champagne-Ardenne
Brief Title: SERUR: COVID-19 Serological Survey of Staff From the University Reims-Champagne Ardennes
Acronym: SERUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-004-SERUR
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID-19; SARS-CoV2 antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population (Experimental): Voluntary people over 18 from the staff of the University of Reims Champagne Ardenne
  Interventions: Diagnostic Test: Anti-SARS-CoV2 Serology

INTERVENTIONS:
Diagnostic Test: Anti-SARS-CoV2 Serology — Diagnostic Test: Anti-SARS-CoV2 Serology A blood sample is collected by venipuncture at Day 0. The anti-SARS-CoV2 serological status is measured by with fully automated MAGLUMI 2019-nCoV IgG and IgM chemiluminescence immunoassays (EUROBIO®)
  Other: Questionnaire
  Data concerning personal exposure factors are collected in a questionnaire:
  * Socio-demographic factors: sex, age,
  * known risk-factor for Covid-19
  * Professional factors: Employment (type, work time, location), protective measures put in place to reduce the risk of contamination
  * Non-professional factors: Contact with infected individuals, carrying of protective equipment and compliance with barrier measures, transport and accomodation modalities during holidays
  Other Names: other : questionnaire

SUMMARY:
This study was designed to determine, in a screening situation within the framework of university preventive medicine, the prevalence of positive anti-SARS-Cov 2 serology among the staff of the University of Reims Champagne-Ardenne. The serological tests chosen will allow systematic detection of anti-SARS-CoV-2 IgM and anti-SARS-Cov-2 IgG to assess the moment of potential contamination prior to resumption of occupational activity.

DETAILED DESCRIPTION:
Objective:

This study was designed to determine, in a screening situation within the framework of university preventive medicine, the prevalence of positive anti-SARS-Cov 2 serology among the staff of the University of Reims Champagne-Ardenne. The serological tests chosen will allow systematic detection of anti-SARS-CoV-2 IgM and anti-SARS-Cov-2 IgG to assess the moment of potential contamination prior to resumption of occupational activity.

Type of study:

This is a prevalence study, a single-center cross-sectional study published on the human person.

Population:

Inclusion criteria: On a voluntary basis, the staff of the University of Reims Champagne Ardenne will be offered a serological blood test (1 dry tube of 7ml). The use of the collected data for research purposes will be explained to each requester, with signature of an informed consent. Only people over 18 will be included.

Non-inclusion criteria: Staff of the University of Reims Champagne Ardenne who have not requested to be tested. Duration of participation of subjects: 1/2 day time

Judgment criterion (s):

Main endpoint (in connection with the main objective): Prevalence of positive SARS-CoV-2 serology at the University of Reims Champagne-Ardenne.

Clinical investigation plan:

* Phase 1: Communication strategy An email will be sent to all the staff of the University of Reims Champagne Ardenne to offer them anti-SARS-Cov-2 serological tests, as part of a health research protocol. Before sampling, a questionnaire will be completed by the applicant.
* Phase 2: Analysis of the samples
* Phase 3: Transmission of results to Pr Frédéric Deschamps, head of SUMMPS at the University of Reims Champagne Ardenne

ELIGIBILITY:
Inclusion Criteria:

* Major volunteers from the Staff of the University of Reims Champagne-Ardenne (>18 years old)

Exclusion Criteria (Non Inclusion):

* persons who do not desire to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of IgG and IgM anti-SARS CoV2 antibodies | Inclusion time was ½ day, time for blood sampling
  Anti-SARS-Cov2 seroprevalence measured in blood sample collected at Day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine GIUSTI, MCU-PH, Principal Investigator — Université de Reims CHampahne-Ardenne - CHU de Reims
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France